CLINICAL TRIAL: NCT02167490
Title: A Randomized Trial Comparing Sentinel Lymph Node Biopsy Vs no Axillary Surgical Staging in Patients With Small Breast Cancer and a Negative Preoperative Axillary Assessment (IEO S637/311)
Brief Title: Sentinel Node Vs Observation After Axillary Ultra-souND
Acronym: SOUND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEO S637/311
Record Dates: First submitted 2014-04-18; First posted 2014-06-19 (Estimated); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Early Stage Breast Carcinoma
Keywords: BC; conservative surgery; SNB; AD; axillary US imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: sentinel node biopsy (Active Comparator): Sentinel node biopsy policy
  Interventions: Procedure: Arm 1: sentinel node biopsy
- Arm 2: observation (No Intervention): No axillary staging

INTERVENTIONS:
Procedure: Arm 1: sentinel node biopsy — Sentinel node biopsy policy
  Arms: Arm 1: sentinel node biopsy

SUMMARY:
The hypothesis of this trial are that:

* avoiding axillary surgery does not worsen the outcome of patients with small breast cancer the absence of the pathological information on the risk of recurrence given by nodal status is not worsening outcome of these patients
* pre-operative imaging of the axilla can identify patients with clinically relevant nodal burden.

The aims of this prospective randomized study are:

* to verify whether, in presence of a negative preoperative axillary assessment, SLN can be spared
* to verify whether, in presence of a negative preoperative axillary assessment, the decision on adjuvant medical treatment can be taken according only to the biology of the tumour without the prognostic information achieved by SLNB on the nodal status
* to verify whether, in presence of a negative preoperative axillary assessment, the patients' quality of life can be improved by a less invasive surgical procedure.

DETAILED DESCRIPTION:
Sentinel lymph node biopsy (SLNB) is the standard approach for axillary staging in patients with breast cancer worldwide. The evident trend of breast cancer treatment is going towards minimizing axillary surgery, even in presence of involvement of the sentinel lymph node (SLN). In fact, it is well known that removal of lymph nodes is performed with staging purposes and to improve regional control but not with curative intent. Recent data from a prospective randomized trial which compared axillary dissection vs. no further axillary surgery in presence of positive SLN did not show any difference in term of overall and disease-free survival. Moreover, to date the impact of the prognostic information of axillary lymph node status in the decision-making process is less important than in the past as the adjuvant treatment is more and more tailored on the biological features of the disease rather than on the risk of recurrence.

This is a prospective randomized controlled trial in which patients with small breast cancer (T<2 cm), with a negative preoperative assessment of the axilla (ultra-sound with FNAC in presence of doubtful findings) will be randomized into two treatment arms:

* SLNB ± axillary dissection
* No axillary surgical staging In the arm 1, no axillary dissection will be performed in case of either negative SLN or in presence of isolated tumour cells or micrometastases. SLNB will be completed by axillary dissection in presence of macrometastases diagnosed in the SLN.

The aims of this prospective randomized study are:

to verify whether, in presence of a negative preoperative axillary assessment, SLN can be spared to verify whether, in presence of a negative preoperative axillary assessment, the decision on adjuvant medical treatment can be taken according only to the biology of the tumour without the prognostic information achieved by SLNB on the nodal status to verify whether, in presence of a negative preoperative axillary assessment, the patients' quality of life can be improved by a less invasive surgical procedure.

Endpoints

The primary endpoint of the study is distant-disease free survival. This endpoint, a proxi of overall survival, will allow to have reliable results in a shorter period of time compared to overall survival.

Secondary endpoints will be the cumulative incidence of distant recurrences, the cumulative incidence of axillary recurrences, the disease free survival (DFS) and the overall survival (OS). Other secondary endpoints are quality of life and evaluation of type of adjuvant treatment administered.

Sample size calculation and statistical considerations

We will consider women who will undergo SLNB as the reference group, and we will test for non-inferiority the group of women not undergoing any treatment in the axilla. For the purpose of sample size calculation, the 5-year DDFS in the reference group is assumed to be 96.5%. Overall, 1560 women (780 per arm) will be enrolled to decide whether the group without treatment of the axilla is no worse than the reference group, given a margin delta of non-inferiority of 2.5% (maximum tolerable 5-years DDFS = 94%). Statistical power and one-sided type I error are set to 80% and 5%, respectively. After 3 years from the start of accrual an interim safety analysis will be performed.

Standard survival analyses and survival analyses with competing events will be performed. Multivariable Cox regression models will be applied to adjust the risk estimates of interest for other variables. The Chi-square test for trend, Chi-square test and the Fisher exact test will be used to evaluate differences in percentages between the two treatment groups, as appropriate. The T-tests will be used to evaluate differences in means for continuous variables.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer <2 cm, and a clinically negative axilla
* any age
* candidates to receive breast conserving surgery + radiotherapy
* negative preoperative assessment of the axilla (ultra-sound with or without FNAC in case one doubtful node is found)
* written informed consent must be signed and dated by the patient and the investigator prior to inclusion.
* patients must be accessible for follow-up.

Exclusion Criteria:

* synchronous distant metastases
* previous malignancy
* bilateral breast cancer
* multicentric or multifocal breast cancer
* previous primary systemic therapy
* pregnancy or breastfeeding
* pre-operative diagnosis (cytology or histology) of axillary lymph node metastases
* pre-operative radiological evidence of multiple involved or suspicious nodes
* patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Distant-disease free survival | 6 months

SECONDARY OUTCOMES:
Cumulative incidence of distant recurrences | 6 months
Cumulative incidence of axillary recurrences | 6 months
Disease free survival (DFS) | 6 months
Overall survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Oreste D Gentilini, MD, Principal Investigator — European Institute of Oncology
Locations (18):
- Instituto Oncologico Fundacion Arturo Lopez Perez, Santiago, Chile
- Italy (15):
  - Comprensorio Sanitario, Bolzano
  - Azienda Ospedaliera Spedali Civili, Brescia
  - Ospedale Oncologico Regionale, Cagliari
  - Humanitas Mater Domini, Castellanza
  - Ospedale S. Anna, Como
  - Azienda Ospedaliera Carlo Poma, Mantova
  - European Institute of Oncology, Milan
  - Fondazione IRCCS Istituto Nazionale Tumori, Milan
  - AOU Federico II, Napoli
  - Istituto Nazionale Tumori, Napoli
  - Ospedale San Matteo, Pavia
  - Ospedale Guglielmo di Saliceto, Piacenza
  - Ospedale Fatebenefratelli, Roma
  - Humanitas Cancer Center, Rozzano
  - Ospedale S. Anna, Torino
- Health Research Institute Hospital La Fe, Valencia, Spain
- Universitätsspital Bern Klinik und Poliklinik für Medizinische Onkologie, Bern, Switzerland

REFERENCES:
- [Background] Veronesi U, Paganelli G, Viale G, Luini A, Zurrida S, Galimberti V, Intra M, Veronesi P, Robertson C, Maisonneuve P, Renne G, De Cicco C, De Lucia F, Gennari R. A randomized comparison of sentinel-node biopsy with routine axillary dissection in breast cancer. N Engl J Med. 2003 Aug 7;349(6):546-53. doi: 10.1056/NEJMoa012782. PMID 12904519
- [Background] Veronesi U, Galimberti V, Paganelli G, Maisonneuve P, Viale G, Orecchia R, Luini A, Intra M, Veronesi P, Caldarella P, Renne G, Rotmensz N, Sangalli C, De Brito Lima L, Tullii M, Zurrida S. Axillary metastases in breast cancer patients with negative sentinel nodes: a follow-up of 3548 cases. Eur J Cancer. 2009 May;45(8):1381-8. doi: 10.1016/j.ejca.2008.11.041. Epub 2009 Jan 6. PMID 19128957
- [Background] Wasif N, Maggard MA, Ko CY, Giuliano AE. Underuse of axillary dissection for the management of sentinel node micrometastases in breast cancer. Arch Surg. 2010 Feb;145(2):161-6. doi: 10.1001/archsurg.2009.269. PMID 20157084
- [Background] Galimberti V, Botteri E, Chifu C, Gentilini O, Luini A, Intra M, Baratella P, Sargenti M, Zurrida S, Veronesi P, Rotmensz N, Viale G, Sonzogni A, Colleoni M, Veronesi U. Can we avoid axillary dissection in the micrometastatic sentinel node in breast cancer? Breast Cancer Res Treat. 2012 Feb;131(3):819-25. doi: 10.1007/s10549-011-1486-2. Epub 2011 Apr 6. PMID 21468637
- [Background] Giuliano AE, McCall L, Beitsch P, Whitworth PW, Blumencranz P, Leitch AM, Saha S, Hunt KK, Morrow M, Ballman K. Locoregional recurrence after sentinel lymph node dissection with or without axillary dissection in patients with sentinel lymph node metastases: the American College of Surgeons Oncology Group Z0011 randomized trial. Ann Surg. 2010 Sep;252(3):426-32; discussion 432-3. doi: 10.1097/SLA.0b013e3181f08f32. PMID 20739842
- [Background] Giuliano AE, Hunt KK, Ballman KV, Beitsch PD, Whitworth PW, Blumencranz PW, Leitch AM, Saha S, McCall LM, Morrow M. Axillary dissection vs no axillary dissection in women with invasive breast cancer and sentinel node metastasis: a randomized clinical trial. JAMA. 2011 Feb 9;305(6):569-75. doi: 10.1001/jama.2011.90. PMID 21304082
- [Background] Fisher B, Jeong JH, Anderson S, Bryant J, Fisher ER, Wolmark N. Twenty-five-year follow-up of a randomized trial comparing radical mastectomy, total mastectomy, and total mastectomy followed by irradiation. N Engl J Med. 2002 Aug 22;347(8):567-75. doi: 10.1056/NEJMoa020128. PMID 12192016
- [Background] International Breast Cancer Study Group; Rudenstam CM, Zahrieh D, Forbes JF, Crivellari D, Holmberg SB, Rey P, Dent D, Campbell I, Bernhard J, Price KN, Castiglione-Gertsch M, Goldhirsch A, Gelber RD, Coates AS. Randomized trial comparing axillary clearance versus no axillary clearance in older patients with breast cancer: first results of International Breast Cancer Study Group Trial 10-93. J Clin Oncol. 2006 Jan 20;24(3):337-44. doi: 10.1200/JCO.2005.01.5784. Epub 2005 Dec 12. PMID 16344321
- [Background] Veronesi U, Orecchia R, Zurrida S, Galimberti V, Luini A, Veronesi P, Gatti G, D'Aiuto G, Cataliotti L, Paolucci R, Piccolo P, Massaioli N, Sismondi P, Rulli A, Lo Sardo F, Recalcati A, Terribile D, Acerbi A, Rotmensz N, Maisonneuve P. Avoiding axillary dissection in breast cancer surgery: a randomized trial to assess the role of axillary radiotherapy. Ann Oncol. 2005 Mar;16(3):383-8. doi: 10.1093/annonc/mdi089. Epub 2005 Jan 24. PMID 15668261
- [Background] Goldhirsch A, Ingle JN, Gelber RD, Coates AS, Thurlimann B, Senn HJ; Panel members. Thresholds for therapies: highlights of the St Gallen International Expert Consensus on the primary therapy of early breast cancer 2009. Ann Oncol. 2009 Aug;20(8):1319-29. doi: 10.1093/annonc/mdp322. Epub 2009 Jun 17. PMID 19535820
- [Background] Colleoni M, Rotmensz N, Peruzzotti G, Maisonneuve P, Mazzarol G, Pruneri G, Luini A, Intra M, Veronesi P, Galimberti V, Torrisi R, Cardillo A, Goldhirsch A, Viale G. Size of breast cancer metastases in axillary lymph nodes: clinical relevance of minimal lymph node involvement. J Clin Oncol. 2005 Mar 1;23(7):1379-89. doi: 10.1200/JCO.2005.07.094. PMID 15735114
- [Background] Montagna E, Viale G, Rotmensz N, Maisonneuve P, Galimberti V, Luini A, Intra M, Veronesi P, Mazzarol G, Pruneri G, Renne G, Torrisi R, Cardillo A, Cancello G, Goldhirsch A, Colleoni M. Minimal axillary lymph node involvement in breast cancer has different prognostic implications according to the staging procedure. Breast Cancer Res Treat. 2009 Nov;118(2):385-94. doi: 10.1007/s10549-009-0446-6. Epub 2009 Jun 27. PMID 19562480
- [Background] Hansen NM, Grube B, Ye X, Turner RR, Brenner RJ, Sim MS, Giuliano AE. Impact of micrometastases in the sentinel node of patients with invasive breast cancer. J Clin Oncol. 2009 Oct 1;27(28):4679-84. doi: 10.1200/JCO.2008.19.0686. Epub 2009 Aug 31. PMID 19720928
- [Background] Korn EL, Hunsberger S, Freidlin B, Smith MA, Abrams JS. Preliminary data release for randomized clinical trials of noninferiority: a new proposal. J Clin Oncol. 2005 Aug 20;23(24):5831-6. doi: 10.1200/JCO.2005.02.105. Epub 2005 Jul 18. PMID 16027441
- [Background] Marubini E, Valsecchi MG. Analysing survival data from clinical trials and observational studies. Chichester, England: Wiley; 1995. 331 pp.
- [Background] Gray RJ. A class of K-sample tests for comparing the cumulative incidence of a competing risk. Ann Statist 1988; 16: 1141-1154
- [Background] Jung SH, Kang SJ, McCall LM, Blumenstein B. Sample size computation for two-sample noninferiority log-rank test. J Biopharm Stat. 2005;15(6):969-79. doi: 10.1080/10543400500265736. PMID 16279355
- [Derived] Gentilini OD, Botteri E, Sangalli C, Galimberti V, Porpiglia M, Agresti R, Luini A, Viale G, Cassano E, Peradze N, Toesca A, Massari G, Sacchini V, Munzone E, Leonardi MC, Cattadori F, Di Micco R, Esposito E, Sgarella A, Cattaneo S, Busani M, Dessena M, Bianchi A, Cretella E, Ripoll Orts F, Mueller M, Tinterri C, Chahuan Manzur BJ, Benedetto C, Veronesi P; SOUND Trial Group. Sentinel Lymph Node Biopsy vs No Axillary Surgery in Patients With Small Breast Cancer and Negative Results on Ultrasonography of Axillary Lymph Nodes: The SOUND Randomized Clinical Trial. JAMA Oncol. 2023 Nov 1;9(11):1557-1564. doi: 10.1001/jamaoncol.2023.3759. PMID 37733364